CLINICAL TRIAL: NCT06403150
Title: The Efficacy and Safety of Levetiracetam Versus Fosphenytoin in Convulsive Status Epilepticus: An Open Label Clinical Trial in Dhaka Medical College Hospital
Brief Title: The Efficacy and Safety of Levetiracetam Versus Fosphenytoin in Convulsive Status Epilepticus
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Dr. Reaz Mahmud, Assistant Professor, Dhaka Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC-DMC/ECC/2023/131
Record Dates: First submitted 2024-02-21; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Status Epilepticus
Keywords: Status Epilepticus; Levetiracetam; Fosphenytoin
MeSH Terms: conditions — Status Epilepticus | interventions — Levetiracetam; fosphenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levetiracetam (Active Comparator): Levetiracetam at 60 mg/kg (max dose 4500 mg) will be intravenously administered in 100mL of normal saline at an administration rate of 2-5mg/kg/min or over 10 minutes.
  Interventions: Drug: Levetiracetam Injection
- Fosphenytoin (Active Comparator): Fosphenytoin at 20 mg/kg (Phenytoin equivalent dose of 15 mg/kg) will be intravenously administered in 100mL of normal saline at an administration rate not exceeding 3mg/kg/min or 150 mg/min.
  Interventions: Drug: Fosphenytoin Injection

INTERVENTIONS:
Drug: Levetiracetam Injection — Levetiracetam at 60 mg/kg (max dose 4500 mg) will be intravenously administered in 100mL of normal saline at an administration rate of 2-5mg/kg/min or over 10 minutes. After 30 minutes following Levetiracetam needle time reassessment of the patient will be done to determine the outcomes.
  Other Names: Iracet Injection; Neurocet Injection
  Arms: Levetiracetam
Drug: Fosphenytoin Injection — Fosphenytoin at 20 mg/kg (Phenytoin equivalent dose of 15 mg/kg) will be intravenously administered in 100mL of normal saline at an administration rate not exceeding 3mg/kg/min or 150 mg/min. After 30 minutes following the Fosphenytoin needle time reassessment of the patient will be done to determine the outcomes.
  Other Names: Fosfen Injection
  Arms: Fosphenytoin

SUMMARY:
Status epilepticus (SE) is an emergency, life-threatening medical condition that may cause irreversible cerebral damage. Therefore, the rapid and secure cessation of seizures and resuscitation is crucial. Potent gamma-aminobutyric acid agonists, including benzodiazepines, are recommended as first-line treatments. For the complete cessation of SE and prevention of recurrence, long-acting antiepileptic drugs (e.g.- FPHT) are also required as second-line treatments along with short-acting benzodiazepines. Intravenous fosphenytoin (FPHT) is associated with fewer adverse events such as life-threatening arrhythmia, cardiac arrest, hypotension, and allergic reactions. Levetiracetam (LEV), is considered to be effective for SE with less serious adverse events including dizziness, somnolence, headache, and transient agitation, but there have been no reports of arrhythmias, hypotension, Stevens-Johnson syndrome, or hepatotoxicity. Preceding studies show that levetiracetam is similarly effective and associated with fewer adverse effects than those of fosphenytoin. Few trials have compared the effectiveness and safety of levetiracetam (LEV) and fosphenytoin (FHP) for status epilepticus worldwide. Moreover, genetic variation is likely to play a crucial role in the development of adverse drug reactions (ADRs) including drug resistance. By far, no study has yet been conducted addressing the issue of efficacy and safety between levetiracetam (LEV) and fosphenytoin (FHP) in status epilepticus in the context of the Bangladeshi population. A comparative study of the efficacy and safety of levetiracetam (LEV) and fosphenytoin (FHP) will be expected to give more confidence for the use of the drug. Considering this the study aims to assess the safety and efficacy of levetiracetam (LEV) and fosphenytoin (FHP) in status epilepticus. This study finding has an implication in the treatment protocol which will be beneficial for the patients and physicians as well. Furthermore, it will give input to the policymaker for developing new guidelines regarding status epilepticus management and also encourage future research.

DETAILED DESCRIPTION:
A randomized control trial will be conducted in the Department of Neurology, DMCH. Ethical approval will be obtained from the DMCH ethical review board before the study. After the selection of the subjects, the nature, purpose, and benefit of the study will be explained to each subject & their legal attendants in detail. They will be encouraged for voluntary participation. Informed written consent will be taken from the participants or their legal attendants. Diagnosis of Status epilepticus will be made according to the criteria of the ILAE task force on classification of status epilepticus (2015). The history of previous disease and habits as well as demographics, the type of SE, seizure duration before treatment, the cause of SE and family history will be recorded. In both groups, height and body weight were estimated from body habitus, family information, or patient records. Blood pressure will be measured. BMI will be calculated as weight (kg)height (m)2. In all patients, neurological assessment will be conducted routinely. Randomized sampling methods will be applied for selecting study subjects. Randomization will be carried out into two groups. After that group A will be treated with FHP and group B will be treated with LEV. Resuscitation and stabilization will be simultaneously performed to ensure airway patency, oxygen inhalation to prevent cerebral hypoxia, securing intravenous access & maintenance of blood pressure. Routine laboratory investigations (full blood count, blood glucose, electrolytes, calcium, magnesium, liver function test & renal function test) will be done. EEG will be done in all patients.

At first, Diazepam will be intravenously administered at 10 mg to all patients. Then, if SE (Status Epilepticus) is not controlled within 20 minutes from Diazepam needle time, study participants will be rapidly randomized and allocated to the FPHT and LEV groups.

In the FPHT group, FPHT at 20 mg/kg (Phenytoin equivalent dose of 15 mg/kg) will be intravenously administered in 100mL of normal saline at an administration rate not exceeding 3mg/kg/min or 150 mg/min.

In the LEV group, LEV at 60 mg/kg (max dose 4500 mg) will be intravenously administered in 100mL of normal saline at an administration rate of 2-5mg/kg/min or over 10 minutes.

Then, after 30 minutes following FPHT/LEV needle time reassessment of the patient will be done to determine the outcomes.

If seizures continue after 30 minutes following FPHT/LEV needle time then, other injectable agents ( e.g- if FPHT given previously, can give LEV intravenously at 60 mg/kg [max dose 4500 mg] or if LEV given previously, can give FPHT intravenously at 20 mg/kg [Phenytoin equivalent dose of 15 mg/kg] ) will be given to the patient.

If seizures still continue after 30 minutes patient will be transferred to intensive care and the standard of care will be given according to intensive care unit protocol.

Once status controlled commence maintenance therapy with Levetiracetam 1000-1500 mg IV twice daily in case of Group-A patient or with FPHT 400 mg/day IV in case of Group-B patient. Subsequent anti-seizure medications will be given based on seizure semiology, etiology, electroencephalography (EEG) correlates, and age of the patient.

After the cessation of seizures, electroencephalography (EEG), neuroimaging (CT / MRI brain), CSF study & other necessary investigations will be performed as needed. FPHT or LEV will be randomized only for the first administration after diazepam and their subsequent administration will be not regulated. The primary outcome will be the seizure cessation rate within 30 minutes of starting administration of the study drug. Secondary outcomes will be the seizure recurrence rate within 24 hours, which will be confirmed by an apparent seizure or non-convulsive seizure detected by EEG; the serious adverse event rate throughout the observational period potentially induced by the study drugs, such as cardiac arrest, life-threatening arrhythmia, respiratory arrest and hypotension and the intubation rate within 24hours. All the information will be recorded in a structured data collection sheet.

Patients will be followed up at 30 minutes, 24 hours, and at discharge after receiving medication and the following outcomes will be assessed: seizure cessation rate, seizure recurrence rate, intubation rate, all-cause in-hospital mortality, adverse effects of drugs, and mRS at discharge. All data will be collected, tabulated, and analyzed statistically using a personal computer and the Statistical Package for Social Science (SPSS) version 26 (IBM, Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with convulsive status epilepticus
* Both male and female
* Willing to give consent

Exclusion Criteria:

* Patients with convulsive status epilepticus already intubated before treatment
* Acute precipitant of seizure was major trauma, hypoglycemia, hyperglycemia, cardiac arrest, or post-anoxia
* Known allergic to FPHT or LEV
* Pregnant patient
* Liver disease or severe renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy and safety between Levetiracetam and Fosphenytoin in adult convulsive status epilepticus. | At 24 hours
  The measurement of a medicine desire effect under ideal conditions, such as clinical trial ( European medicine agency). It is measured as percentage in reduction of seizure frequency from the time of drug initiation and also measure the Incidence of treatment-emergent adverse events.

SECONDARY OUTCOMES:
Seizure cessation rate | Thirty minutes
  Seizure cessation rate was calculated by the ratio between number of patients admitted with status epilepticus and number of patient free from convulsion after administration of intervention drug
Seizure recurrence rate within 24 hours | 24 hours
  seizure recurrence rate within 24 hours, which was confirmed by an apparent seizure or non-convulsive seizure detected by EEG
Observe and compare the serious adverse event rate | At 30 minutes, at 24 hours and at Hospital discharge
  Any noxious, unintended and undesired effect (including an abnormal laboratory finding) of a drug which occurs at a dose used in humans for prophylactic, diagnostic or therapeutic purpose (WHO)
Intubation rate within 24hours | 24 hours
  Patient need intubation and mechanical ventilation
All-cause in-hospital mortality among patients | From date of randomization until the date of death from any cause
  Death during hospital admission period from all causes
Modified Rankin Scale (mRS) score | At 30 minutes, at 24 hours and at Hospital discharge
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. mRS score '0' means patient has no residual symptoms and score '6' means patient has expired

CONTACTS AND LOCATIONS:
Overall Officials: Dr Md Amirul Islam, MBBS, Principal Investigator — MD (Neurology) Phase B Resident; Professor Dr Kazi Gias Uddin Ahmed, MD, Study Chair — Professor of Neurology, Dhaka Medical College; Dr Reaz Mahmud, MD, Study Director — Assistant Professor of Neurology, Dhaka Medical College
Locations (1):
- Dhaka Medical College Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Demographic variables, Primary and Secondary outcomes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: May 2023 to October 2024
Access Criteria: Those who works with Status Epilepticus patients